CLINICAL TRIAL: NCT01149681
Title: Open-label, Phase II Clinical Trial of Aplidin® (Plitidepsin) in Patients With Primary Myelofibrosis (PMF) and Post Polycythemia Vera/Essential Thrombocythemia (Post-PV/ET) Myelofibrosis
Brief Title: Clinical Trial of Aplidin® in Patients With Primary Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL-B-020-10
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: Myelofibrosis
Keywords: Aplidin; Plitidepsin; Myelofibrosis; Pharma Mar
MeSH Terms: conditions — Primary Myelofibrosis | interventions — plitidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm one (Experimental)
  Interventions: Drug: APLIDIN (plitidepsin)

INTERVENTIONS:
Drug: APLIDIN (plitidepsin) — Aplidin® (plitidepsin) lyophilized powder and solvent for concentrate for solution for infusion. (2 mg plitidepsin vial and 4 ml ampoule).
  Plitidepsin will be administered at 5 mg/m2 intravenously diluted to a total volume of 250 ml in 0.9% saline or 5% dextrose solution on Day 1 and 15 every four weeks for a maximum period of 6 cycles.

SUMMARY:
This is an open-label, Phase II Clinical Trial of Aplidin® (plitidepsin) in Patients with Primary Myelofibrosis and post polycythemia vera/essential thrombocythemia (Post-PV/ET) Myelofibrosis.

DETAILED DESCRIPTION:
This trial tries to assess response rate (ORR) of plitidepsin in patients with:

primary myelofibrosis (PMF), post-polycythemia vera myelofibrosis (post-PV MF), or post-essential thrombocythemia myelofibrosis (post-ET MF). Besides, the study results will allow to evaluate the effect of plitidepsin on bone marrow (BM) or peripheral blood histology and to determine the quality of life (QoL) and symptoms or participant patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Primary Myelofibrosis (PMF) or Post Polycythemia Vera/Essential Thrombocythemia Myelofibrosis(post-ET/PV MF) as per revised World Health Organization (WHO) criteria.
2. High-risk or intermediate-2 risk Myelofibrosis (MF) as defined by the International Prognostic Scoring System (IPSS); or intermediate-I risk MF associated with symptomatic splenomegaly/hepatomegaly and/or unresponsive to available therapy.
3. At least 18 years of age, with life expectancy of ≥12 weeks.
4. Able to provide informed consent and being willing to sign an informed consent form (ICF).
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
6. Evidence of acceptable organ function within seven days of initiating study drug

Exclusion Criteria:

1. Previous treatment with plitidepsin.
2. Any of the following therapies within two weeks prior to initiation of study drug:

   * chemotherapy (e.g., hydroxyurea),
   * immunomodulatory drug therapy (e.g., thalidomide),
   * immunosuppressive therapy,
   * corticosteroids >10 mg/day prednisone or equivalent, or
   * erythropoietin.
3. Incomplete recovery from major surgery within four weeks of study entry.
4. Radiation therapy within four weeks of study entry.
5. Women of childbearing potential
6. Women who are pregnant or are currently breastfeeding.
7. Myopathy grade > 2
8. Known positive status for human immunodeficiency virus (HIV).
9. Active hepatitis B or C virus (HBV or HCV) infection
10. Diagnosis of another invasive malignancy
11. Any acute active infection.
12. Known hypersensitivity to the study drug or any of its formulation components (e.g., Cremophor®).
13. Treatment with any investigational product in the 30 days before inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- Azienda Ospedaliero Universitaria Careggi di Firenze, Florence, Italy

RESULTS

PARTICIPANT FLOW:
Groups:
- Aplidin®: APLIDIN (plitidepsin): Aplidin® (plitidepsin) lyophilized powder and solvent for concentrate for solution for infusion. (2 mg plitidepsin vial and 4 ml ampoule).
  Plitidepsin will be administered at 5 mg/m2 intravenously diluted to a total volume of 250 ml in 0.9% saline or 5% dextrose solution on Day 1 and 15 every four weeks for a maximum period of 6 cycles.
Period: Overall Study
Arm/Group | Aplidin®
Started | 12
Completed | 0
Not Completed | 12
Not completed — Withdrawal by Subject | 7
Not completed — Progressive disease | 1
Not completed — Physician Decision | 2
Not completed — adverse events nonrelated study drug | 2

BASELINE CHARACTERISTICS:
Arm/Group | Aplidin®
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10
  Italy | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) of plitidepsin in patients with: primary myelofibrosis (PMF), post-polycythemia vera myelofibrosis or post-essential thrombocythemia myelofibrosis.
  ORR according to the International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) response criteria (Tefferi et al., 2006) in the evaluable population: defined as a confirmed disease response, on two consecutive evaluations performed at least eight weeks apart. Overall response (OR) = Complete Response (CR) + Partial response (PR) + Clinical improvement (CI).
Time Frame: All patients were followed up to progressive disease, start of a new anti-cancer therapy, death or one year after the last treatment visit of the last patient, whichever occured first
Population: 1 of the 12 patients treated was excluded. This patient received 1 complete infusion of plitidepsin in Cycle 1, and had the second infusion interrupted due to plitidepsin-related grade 3 chest and epigastric pain (reported as SAEs). Although the episode resolved a day later, she refused to continue treatment and had no disease evaluations done
Measure: Count of Participants; unit: Participants
Arm/Group | Arm One
Number analyzed (Participants) | 11
Participants
  Clinical improvement | 1
  Stable disease | 9
  Progressive disease | 1

2. Secondary Outcome: Quality of Life (QoL)
Description: Quality of life (QoL) and symptoms assessment according to the Myelofibrosis Symptom Assessment Form (MFSAF), after treatment with plitidepsin. For full details please refer to Mesa RA, Schwager S, Radia D, Cheville A, Hussein K, Niblack J, et al. The Myelofibrosis Symptom Assessment Form (MFSAF): an evidence-based brief inventory to measure quality of life and symptomatic response to treatment in myelofibrosis. Leuk Res 2009;33(9):1199-203.
  Scale measures: 0 to 10 (0 if absent) ranking being 1 the most favorable and 10 least favorable.
Time Frame: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aplidin®
Number analyzed (Participants) | 12
score on a scale
  Overall quality of life - Baseline | 5.7 [4.8 to 6.6]
  Overall quality of life - Cycle 1 | 5.0 [4.1 to 5.9]
  Overall quality of life - Cycle 2 | 5.4 [3.8 to 6.9]
  Overall quality of life - Cycle 3 | 6.3 [3.5 to 9.2]
  Overall quality of life - Cycle 4 | 7.5 [-24.3 to 39.3]
Statistical Analysis 1: Comparison: Aplidin®; Test type: Superiority; p = 0.2364, Repeated measures analysis

3. Other Pre Specified Outcome: Progression-free Survival (PFS)
Description: Progression free survival (PFS) is defined as the time from start of treatment to the date of documented progressive disease (PD) by IWG-MRT criteria or death (regardless of the cause of death), whichever comes first. Patients who progress or die will be considered to have had an event, except if this event occurs after the start of subsequent antitumor therapy, in which case the patient will be censored at the time of last disease assessment prior to or on the first day of the first subsequent antitumor therapy. If the patient is lost for the assessment of progression during the follow-up period, or has more than one missing follow-up between the date of last tumor assessment and the date of progression, death or further antitumor therapy, the PFS will be censored at the date of last valid disease assessment before the missing evaluations.
Time Frame: All patients were followed up to progressive disease or death, whichever occured first, up to 30 days after their last dose
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Aplidin®
Number analyzed (Participants) | 11
months | 4.6 [1.4 to 4.6]

ADVERSE EVENTS:
Arm/Group | Aplidin®
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aplidin® (N=12)
Anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Bronchopneumonia (Infections and infestations) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aplidin® (N=12)
Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Aortic valve disease (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus arrhythmia (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 5
Faeces discoloured (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 5
Early satiety (General disorders) | 8
Fatigue (General disorders) | 12
Infusion related reaction (General disorders) | 1
Oedema (General disorders) | 3
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 2
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 3
Electrocardiogram T wave abnormal (Investigations) | 2
Troponin T increased (Investigations) | 1
Weight decreased (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Iron overload (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 6
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Balance disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 2
Haematuria (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash macular (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Pallor (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days